CLINICAL TRIAL: NCT05119231
Title: Pulmonary Vein Isolation Versus SHAM-pulmonary Vein Isolation for Symptomatic Relief in Patients With Atrial Fibrillation- a Randomised Trial - PVI-SHAM-AF
Brief Title: Pulmonary Vein Isolation vs SHAM-pulmonary Vein Isolation for Symptomatic Relief in Patients With AF
Acronym: PVI-SHAM-AF
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Leipzig (Other)
Responsible Party: Principal Investigator, Rolf Wachter, Professor, University of Leipzig
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: PVI-SHAM-AF CIV-21-01-035584
Record Dates: First submitted 2021-11-03; First posted 2021-11-15 (Actual); Last update posted 2025-11-19 (Actual); Status verified 2025-11

CONDITIONS: Atrial Fibrillation
Keywords: Arrhythmias, Cardiac; Heart Disease; ECG Monitoring
MeSH Terms: conditions — Atrial Fibrillation; Arrhythmias, Cardiac; Heart Diseases

STUDY DESIGN:
Intervention Model Description: randomized, parallel group, sham-controlled and double-blinded multicenter trial
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Pulmonary Vein Isolation (Experimental): Pulmonary Vein Isolation (radiofrequency ablation or cryoablation) of atrial fibrillation according to local standards:
  Trial participants will assigned to the PVI-arm will undergo catheter ablation within 48 hours after baseline evaluation, with the aim to achieve isolation of all pulmonary veins and restore sinus rhythm.
  Dependent of the local standards an echocardiography or cardiac MRI will be performed prior to the procedure. If necessary, a transesophageal echocardiography must be performed to exclude presence of atrial thrombus.
  Anticoagulation will be initiated/continued for at least 3 months after the procedure.
  Interventions: Procedure: Pulmonary Vein Isolation
- Sham Control Arm (Sham Comparator): Sham Pulmonary Vein Isolation
  Trial participants will assigned to the SHAM-arm will undergo their procedure within 48 hours after baseline evaluation. The Sham procedure will include deep sedation according to the respective PVI protocol for at least one hour, femoral vein/artery puncture with introduction of sheaths and an electrical cardioversion in presence of persistent atrial fibrillation.
  Dependent of the local standards an echocardiography or cardiac MRI will be performed prior to the procedure. If necessary, a transesophageal echocardiography must be performed to exclude presence of atrial thrombus.
  Anticoagulation will be initiated/continued for at least 3 months after the procedure.
  Interventions: Other: Sham-Pulmonary Vein Isolation

INTERVENTIONS:
Procedure: Pulmonary Vein Isolation — Catheter ablation (radiofrequency ablation or cryoablation) of atrial fibrillation according to local standard
  Arms: Pulmonary Vein Isolation
Other: Sham-Pulmonary Vein Isolation — Sham-Pulmonary Vein Isolation in deep sedation for at least one hour including femoral vein/artery puncture with introduction of sheaths and electrical cardioversion in presence of current atrial fibrillation
  Arms: Sham Control Arm

SUMMARY:
Being the most common arrhythmia, atrial fibrillation (AF) is a high burden of public health with an increasing prevalence in our aging population. Interventional treatment of atrial fibrillation by catheter ablation is one of the treatment pillars in the complex field of "better symptom control" based on current Guidelines. Catheter ablation of atrial fibrillation is based on electrical isolation of the pulmonary veins (pulmonary vein isolation: PVI) from the left atrium. The main benefit and goal of PVI in AF patients is the reduction of AF-related symptoms, resulting in an improvement of quality of life. It was shown, that catheter ablation failed to prove a difference in AF recurrence after PVI compared to medical therapy in the first 18 month of follow-up. It was also shown, that these episodes will become more asymptomatic. This raises concerns that the symptomatic improvement might be the result of a placebo effect, which will be elucidated with this study.

DETAILED DESCRIPTION:
Being the most common arrhythmia, atrial fibrillation (AF) is a high burden of public health with an increasing prevalence in our aging population. Interventional treatment of atrial fibrillation by catheter ablation is one of the treatment pillars in the complex field of "better symptom control" based on current Guidelines. Atrial fibrillation is commonly induced and maintained by abnormal electrical impulses originating in the pulmonary veins. Catheter ablation of atrial fibrillation is based on electrical isolation of the pulmonary veins (pulmonary vein isolation: PVI) from the left atrium. This is achieved either by heating (Radiofrequency ablation) or freezing (Cryoablation) of the tissues. By inducing the formation of scar tissue, the pulmonary veins are "electrically isolated" and abnormal electrical signals are not transferred any more to the left atrium.

The main benefit and goal of PVI in AF patients is the reduction of AF-related symptoms, resulting in an improvement of quality of life. The effect was shown to be significantly higher compared with conventional medical treatment. In contrast, there is no evidence for a substantial effect of PVI on hard clinical endpoints. The recent large randomized controlled trial CABANA (Catheter ABlation vs. ANtiarrhythmic Drug Therapy for Atrial Fibrillation) did not show a reduction of the primary composite endpoint of death, disabling stroke, serious bleeding and cardiac arrest in the intention-to-treat analysis although the results are highly controversial due to the high crossover rate.

Up to now, the only patient population with evidence for a prognostic benefit of PVI in symptomatic AF are patients with a heart failure and a reduced ejection fraction (HFrEF). In the CASTLE-AF trial, a relative risk reduction for all-cause mortality of 47% was shown for HFrEF patients with AF ablation compared with conventional treatment.

7-Day Holter monitoring in patients 6 month after treatment with PVI revealed a significant increase in asymptomatic AF episodes. Furthermore, the MANTRA-PAF randomised trial (Medical Antiarrhythmic Treatment or Radiofrequency Ablation in Paroxysmal Atrial Fibrillation) failed to prove a difference in AF recurrence after PVI compared to medical therapy in the first 18 month of follow-up.

This raises concerns that the symptomatic improvement might be the result of a placebo effect.

PVI-SHAM-AF is a prospective, double-blinded, sham-controlled, randomized, multicenter trial whose aim is to compare the effect of catheter-based ablation on patient reported outcomes based on common AF questionnaires with a sham procedure. 260 patients without previous PVI or surgical treatment of atrial fibrillation, a LVEF >35% and an indication for interventional treatment of AF with pulmonary vein isolation based on current Guidelines (ESC 2020) will be enrolled and randomized 2:1 to undergo either PVI or sham procedure. The latter will include deep sedation as performed during standard PVI treatment for at least one hour, introduction of femoral sheaths and if necessary electrical cardioversion in patients with persisting AF. No catheter will be placed within the participant. The official procedure protocol will include no details about the intervention; postinterventional care will be conducted independent of whether a catheter ablation or sham procedure was performed, based on the respective PVI protocol.

Patient will be followed up for one year with visit at 3, 6 and 12 months. Each of these visits include questionnaires for AF related Symptoms (AFEQT, SF-36 and EQ-5D); 7-Day Holter Monitoring will be performed 6 months after the procedure. Participants will be unblinded after 12 months. The primary endpoint will be the difference of AFEQT sum scores evaluated at 6 months to baseline.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with symptomatic atrial fibrillation scheduled for pulmonary vein isolation
2. Class I or class IIa indication for pulmonary vein isolation by current guidelines
3. Age ≥ 18 years
4. Written informed consent

Exclusion Criteria:

1. History of previous pulmonary vein isolation or surgical treatment of atrial fibrillation
2. Reversible causes of atrial fibrillation (e. g. thyroid disorder, acute alcohol intoxication, recent major surgical procedures, trauma or acute infection)
3. Moderate or severe valvular heart disease
4. CHA2DS2-VASc-Score =0 (males) or 1 (females) or contraindication to oral anticoagulation
5. Acute coronary syndrome, percutaneous coronary intervention, valve surgery or percutaneous intervention or cardiac bypass surgery and stroke within the last 3 months
6. Reduced left ventricular ejection fraction < 35%
7. Hypertrophic obstructive cardiomyopathy
8. Medical conditions limiting the expected survival to < 1 year
9. Participation in any other randomized controlled trial
10. Women of childbearing potential without appropriate contraceptive measures (oral contraceptives, vaginal ring, intrauterine devices, implanon, injections, partner with vasectomy) pregnant woman or woman with desire for children
11. Any condition that - in the opinion of the investigator - may prevent the subject from adhering to the study protocol (e.g. history of non-compliance, drug addiction)
12. Subjects under legal supervision or guardianship
13. Unable to give informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 262 (Actual)
Dates: Start 2021-11-12 (Actual); Primary Completion 2026-05 (Estimated); Study Completion 2026-11 (Estimated)

PRIMARY OUTCOMES:
difference of AFEQT sum scores evaluated at 6 months | 6 months after randomisation compared to baseline
  The primary objective is to show a significant improvement of AF symptoms (measured by AFEQT sum score) by PVI in comparison to sham-PVI, evaluated six months after randomisation compared to baseline.
  Primary endpoint is the difference of AFEQT sum scores between the PVI and the sham-PVI arm, evaluated at 6 months after randomisation.

SECONDARY OUTCOMES:
the longitudinal change of the AFEQT score | baseline - 3, 6 and 12 months
  improvement of AF symptoms (measured by AFEQT sum score) by PVI in comparison to sham-PVI, evaluated at 3, 6 and 12 months after randomisation compared to baseline.
difference of EQ-5D scores | at 6 months to baseline
  improvement of AF symptoms (measured by EQ-5D sum score) by PVI in comparison to sham-PVI, evaluated six months after randomisation compared to baseline.
difference of SF-36 scales | at 6 months to baseline
  improvement of AF symptoms (measured by SF-36 sum score) by PVI in comparison to sham-PVI, evaluated six months after randomisation compared to baseline.
the change of EQ-5D over time (baseline - 3, 6 and 12 months) in a longitudinal view | (baseline - 3, 6 and 12 months) in a longitudinal view
  improvement of AF symptoms (measured by EQ-5D sum score) by PVI in comparison to sham-PVI, evaluated at 3, 6 and 12 months after randomisation compared to baseline.
the change of SF-36 over time | baseline - 3, 6 and 12 months
  improvement of AF symptoms (measured by SF-36 sum score) by PVI in comparison to sham-PVI, evaluated at 3, 6 and 12 months after randomisation compared to baseline.
AF burden measured as percentage of time in AF during 7 day Holter ECG monitoring | at 6 months
  AF burden measured as percentage of time in AF during 7 day Holter ECG monitoring
Incidence of AF recurrence | at 3, 6 and 12 months
  measured by patient reports and external ECGs
N-terminal-proBNP plasma levels | at 6 months
  change of baseline N-terminal-proBNP plasma levels in comparison to 6 months after randomisation

CONTACTS AND LOCATIONS:
Overall Officials: Rolf Wachter, Prof. Dr., Study Chair — University of Leipzig
Locations (9):
- Germany (8):
  - Regiomed Klinikum, Coburg, Bavaria
  - University Hospital Gießen, Giessen, Hesse
  - Universitätsklinikum Münster, Münster, North Rhine-Westphalia
  - Heart Center Dresden University Hospital, Dresden, Saxony
  - German Heart Center of Charité University Medicine, Standort Charité Mitte, Berlin, State of Berlin
  - German Heart Center of Charité University Medicine, Standort DHZB, Berlin, State of Berlin
  - Herzzentrum Leipzig, Leipzig
  - Universitätsklinikum Leipzig, Leipzig
- Department of Cardiology, Silesian Center for Heart Diseases, Zabrze, Poland

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP, ICF
Time Frame: with publication of the major results
Access Criteria: IPD will be made available upon reasonable request and if approved by the ethic´s committee.
URL: https://www.zks.uni-leipzig.de/

REFERENCES:
- [Background] Dilk P, Uhe T, Forkmann M, Eckardt L, Bode K, Seewoster T, Gaspar T, Neef M, Dinov B, Bacak M, Petroff D, Prettin C, Hindricks G, Laufs U, Dagres N, Wachter R. Pulmonary vein isolation versus SHAM-pulmonary vein isolation for symptomatic relief in patients with atrial fibrillation-Design and rationale of the PVI-SHAM-AF trial. Am Heart J. 2025 Dec;290:93-104. doi: 10.1016/j.ahj.2025.06.003. Epub 2025 Jun 11. PMID 40513974